CLINICAL TRIAL: NCT01608035
Title: Ultrasound Guided Sciatic Perineural Catheter vs Surgically Placed Sciatic Stump Catheter for Below Knee Amputations: Is There A Difference in Patient Outcomes
Brief Title: Sciatic Perineural Versus Stump Catheter for Below Knee Amputation
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H12-00693
Record Dates: First submitted 2012-05-11; First posted 2012-05-30 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Ischemia; Phantom Limb Pain; Vascular Disease; Chronic Pain
Keywords: sciatic catheter; stump catheter; below knee amputation
MeSH Terms: conditions — Ischemia; Phantom Limb; Vascular Diseases; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sciatic catheter (Experimental)
  Interventions: Procedure: Sciatic catheter
- Stump catheter (Active Comparator)
  Interventions: Procedure: Stump catheter

INTERVENTIONS:
Procedure: Sciatic catheter — presurgical sciatic catheter insertion
  Other Names: anesthesiologist placed catheter
  Arms: sciatic catheter
Procedure: Stump catheter — intraoperative placed stump catheter
  Other Names: surgeon placed catheter
  Arms: Stump catheter

SUMMARY:
The goal of this study is to determine if pre-operative placement of the continuous peripheral nerve block by an anesthesiologist using ultrasound technology is more effective than a continuous peripheral nerve block placed during the surgery by a surgeon for patients undergoing a limb amputation

DETAILED DESCRIPTION:
We wish to determine the most effective site for the continuous infusion of local anesthetic for patients undergoing amputation of a limb. The information we obtain from this study will help to decide the most effective manner to provide pain relief for patients in the future. The primary outcome of interest is post-operative pain relief as measured by the amount of pain-relieving medications (opioids) required by patients prior to discharge home. The secondary outcomes of interest will be pain-relieving medications (opioid) requirements during the operation, length of stay in the hospital, time required for mobility, and patient satisfaction- measured by a survey given while in hospital and 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* undergoing a below knee amputation
* 16 years of age or older
* regional anesthetic will be used as part of the surgery

Exclusion Criteria:

* pregnant
* allergic to local anesthetic or ultrasound jelly
* a contraindication to having a peripheral nerve block catheter

Ages: 16 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Post-op day 0-7
  MAR records will be used to calculate opioid consumption

SECONDARY OUTCOMES:
pain score | Post-op day 0-7 and at 3months
  VAS will be used (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew N Sawka, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- Jason Wilson, Vancouver, British Columbia, Canada